CLINICAL TRIAL: NCT03661164
Title: Factors Influencing Keratoconus Progression After Iontophoretic Transepithelial Corneal Cross-linking in Pediatric Patients: Three Year Follow up
Brief Title: Iontophoretic Transepithelial Corneal Cross-linking in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Luca Buzzonetti (Other)
Responsible Party: Sponsor-Investigator, Luca Buzzonetti, Head of the Ophthalmology Department, Bambino Gesù IRCCS Children's Hospital, Rome, Italy, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: ICXL
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: corneal cross linking — Iontophoretic corneal cross linking

SUMMARY:
To report three year follow up in pediatric patients with keratoconus after iontophoretic transepithelial corneal cross-linking (CXL) to assess preoperative factors that may influence ectasia progression

DETAILED DESCRIPTION:
Purpose: To report three year follow up in pediatric patients with keratoconus after iontophoretic transepithelial corneal cross-linking (CXL) to assess preoperative factors that may influence ectasia progression.

Methods: Thirthyfive eyes of 22 consecutive pediatric patients (mean age 14.3±2.5 years) with keratoconus are evaluated in this retrospective study. Subgroup A and B are made up in function of progression in maximum K (Kmax,) defined as steepening of 1.0 diopter or more recorded three year after CXL. Corrected distance visual acuity (CDVA), spherical equivalent, topographic cone location, Kmax, posterior elevation of the thinnest point and thinnest point are evaluated. A paired Student t test is used to compare preoperative and 12, 24, and 36 month postoperative da-ta. A P value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of Keratoconus age < 18 years at the treatment iontophoretic corneal cross linking performed at least 3 years before

Exclusion Criteria:

age > 18 years at the treatment

I

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Thirtyfive eyes of 22 consecutive pediatric patients (5 female and 17 male; mean age 14.3±2.5 [SD] years; range, 9 to 18 years) affected by keratoconus (diagnosis established accord-ing to global consensus on keratoconus and ectatic diseases) who underwent transepithelial corneal cross-linking by iontophoresis are enrolled in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
: Preoperative Kmax | 3 years
  Simulated maximum K (Kmax) is calculated by a Sirius Scheimpflug camera (CSO, Firenze, Italy) by averaging the axial curvature from the fourth to the eighth Placido rings of the flattest and steepest meridians (the amplitude of the zone taken into consideration, therefore has a vari-able diameter depending on the curvature of the cornea, and the principal meridians are not nec-essarily 90 degrees away)
posterior elevation of the thinnest point | 3 years
  posterior elevation of the thinnest point is measured by a Sirius Scheimpflug camera (CSO, Firenze, Italy)
cone location | 3 years
  The topographic cone location is assessed at the preoperative visit as follows : central for cor-neas having maximum K located within the central 3 mm and paracentral for corneas having maximum K located within the central 3 to 5 mm.